CLINICAL TRIAL: NCT05606549
Title: Effect of Marital Self Disclosure Intervention on Fear of Cancer Recurrence and Dyadic Coping Ability Among Gastric Cancer Survivors and Their Spouse
Brief Title: Effect of MSD on FCR Among Gastric Cancer Survivors
Acronym: MSD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Malaya (Other)
Collaborators: Jiangsu Taizhou People's Hospital (Other); Jingjiang People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 18801155781
Record Dates: First submitted 2022-10-21; First posted 2022-11-04 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-10

CONDITIONS: Stomach Cancer；Clinical Control Trial
Keywords: Cancer Survivors；Stomach；Marital Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- marital self disclosure (Experimental)
  Interventions: Behavioral: Marital self disclosure
- Routine care (No Intervention)

INTERVENTIONS:
Behavioral: Marital self disclosure — Intervention time during hospitalization is the first day after chemotherapy, and intervene once per chemotherapy, a total of 4 times, 40-60 min each time. Interventions included verbal and written disclosure. The researcher will preside over the MSD process and introduce of MSD for gastric patients and their spouse，both patient and their spouse will receive a training or review on MSD skills, 5-10 minutes each time. Couples practice MSD skills through 4 revealing themes. Couples are encouraged to express their FCR, and when one partner disclosure, supporters should allow the speaker to fully express their feelings and respond positively to the speaker's message, showing empathy for them, and acknowledging their point of view.
  Arms: marital self disclosure

SUMMARY:
The goal of this clinical trial is to explores the effect of marital self disclosure intervention on fear of cancer recurrence and dyadic coping ability in gastric cancer survivors and their spouses. The main questions are: What is the level of fear of cancer recurrence among gastric cancer survivors and their spouse? What is the level of dyadic coping ability among gastric cancer survivors and their spouse?What is the effect of marital self-disclosure intervention on fear of cancer recurrence and dyadic coping ability in the gastric cancer survivors and their spouses? Participants will accept the intervention of marital self disclosure for 4 times (4 cycles of chemotherapy) with different topics. Researchers will compare with control group to see if the level of fear of cancer recurrence and dyadic coping ability will be improved.

ELIGIBILITY:
Inclusion Criteria:

* The disease meets the diagnostic criteria of "Guidelines for Diagnosis and Treatment of Gastric Cancer"(Department of Medical Affairs, 2019), the preoperative gastroscopy and pathological diagnosis are advanced gastric cancer, and the postoperative pathological classification is type II, III or IV
* Age ≥ 18 years
* Able to write and oral communicate effectively by themself
* The main caregiver is their spouse
* Clear consciousness, no understanding barriers
* Agree to participate in this study

Exclusion Criteria:

* History of receiving a structured psychological intervention from a psychiatrist or a psychologist
* Cognitive disorders or psychiatric disorders (according to the DSM-V)
* Severe visual, hearing and speech impairment
* With previous or concurrent malignant tumors
* With severe complications, such as gastrointestinal obstruction, perforation, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2022-10-19 (Actual); Primary Completion 2023-10-25 (Estimated); Study Completion 2024-04-20 (Estimated)

PRIMARY OUTCOMES:
Fear of Progression Questionnaire-Short form (FoP-Q-SF) for Patients | 4 months
  The FoP-Q-SF is a one-dimensional scale constructed by on the basis of the Fear of Progression Questionnaire (FoP-Q). The FoP-Q-SF for Patients scale includes 12 items, using 5-point Likert Scale, 1 point means "never", 5 points means "always", with a total score ranging from 12 to 60, with higher scores indicating higher fear of disease progression.
Fear of Progression Questionnaire-Short form (FoP-Q-SF) for Partners | 4 months
  FoP-Q-SF for Partners is developed by Zimmermann et al. (2011) based on the structure of the FoP-Q-SF scale to assess the degree of disease progression of the patient's spouse's fear of disease. FoP-Q-SF for Partners includes 12 items, adopting 5-point Likert scale, 1 point representing "never" and 5 points representing "always", with a total score ranging from 12 to 60, with higher scores indicating higher fear of their spouse's disease progression.

SECONDARY OUTCOMES:
Dyadic Coping Inventory(DCI) | 4 months
  DCI based on the system interaction model was originally developed by Bodenmann ( 2000), which includes 6 dimensions, 55 items, and use Likert 5-point scale. After further improvement, the DCI (Bodenmann & Randall, 2012) was revised to 37 items and measured on a 5-point Likert scale, ranging from 1 (not at all/very rarely) to 5 (very often).

CONTACTS AND LOCATIONS:
Locations (1):
- Jingjiang people's Hospital, Taizhou, Jiangsu, China

REFERENCES:
- [Derived] Zhao H, Zhou Y, Che CC, Chong MC, Zheng Y, Hou Y, Chen C, Zhu Y. Marital Self-Disclosure Intervention for the Fear of Cancer Recurrence in Chinese Patients With Gastric Cancer: Protocol for a Quasiexperimental Study. JMIR Res Protoc. 2024 Apr 29;13:e55102. doi: 10.2196/55102. PMID 38684089